CLINICAL TRIAL: NCT01299597
Title: A Single-centre Open Label Study to Investigate the Effect of Repeat Doses of SB-649868 on the Pharmacokinetics of Simvastatin and Atorvastatin in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 109652
Record Dates: First submitted 2010-07-01; First posted 2011-02-18 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Sleep Disorders
Keywords: repeat dose; statins; safety and tolerability; drug interaction; sb649868; healthy male subjects; pharmacokinetics
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Atorvastatin; Simvastatin; N-((1-((5-(4-fluorophenyl)-2-methyl-4-thiazolyl)carbonyl)-2-piperidinyl)methyl)-4-benzofurancarboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1: Atorvastatin (Experimental): single dose session with Atorvastatin with PK samples collected up to 72h post dose, then 14 days repeat dose session with SB649868 with Atorvastatin single dose co-administered on day 8 (same time as SB649868) and on day 12 (2 hours before SB649868).
  Interventions: Drug: Atorvastatin; Drug: SB649868
- Cohort 2: Simvastatin (Experimental): single dose session with Simvastatin with PK samples collected up to 24h post dose, then 14 days repeat dose session with SB649868 with Simvastatin single dose co-administered on day 12 (same time as SB649868) and on day 14 (2 hours before SB649868).
  Interventions: Drug: Simvastatin; Drug: SB649868

INTERVENTIONS:
Drug: Atorvastatin — 20mg single dose given alone and coadministered with SB649868 on day 8 and 12 of the 14-day repeat dose period.
  Arms: Cohort 1: Atorvastatin
Drug: Simvastatin — 10mg single dose given alone and coadministered with SB649868 on day 12 and 14 of the 14-day repeat dose period.
  Arms: Cohort 2: Simvastatin
Drug: SB649868 — 20mg daily given for 14 days.

SUMMARY:
The present study will investigate in humans the enzyme inhibition effects of SB-649868 on CYP3A4, using Simvastatin and Atorvastatin as CYP3A4 probe substrates, administered as single doses: alone, and on two different occasions after repeat doses of SB-649868, at the same time as SB-649868 and 2h before SB-649868.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subject, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, neuropsychiatric status using the MINI International Neuropsychiatric Interview, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. However,

   * Subjects with cTpn I values above 99th percentile of normal range of the selected assay should always be excluded from enrollment;
   * Subjects with alkaline phosphatase or bilirubin > 1.5xULN should always be excluded (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%);
2. Male between 18 and 65 years of age inclusive, at the time of signing the informed consent.
3. Body weight ≥50 kg and BMI within the range 18.5-29.9 kg/m2 inclusive.
4. Subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 3 days post last dose (equivalent to 5 terminal half-lives post-last dose).
5. Having given written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

1. History or presence of significant psychiatric neurological, musculo-skeletal , respiratory, gastrointestinal, hepatic, uncontrolled hypothyroidism. pancreatic or renal diseases or of any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
2. Subjects, who in the Investigator's judgement, pose a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behaviour and/or any suicidal ideation of type 4 or 5 on the C-SSRS in the last 6 months.
3. History of cardiovascular diseases and/or evidence of repolarization defects.
4. Family history of heriditary muscular disorders.
5. Subjects with abnormal ECG defined as: average QTcB or QTcF > 450 msec; PQ < 120 ms or > 220 ms; complete left bundle branch block; second-or third-degree AV block; any relevant ST/T wave abnormalities ; any atrial or ventricular arrhtymias which are of clinical significance as determined by the Investigator.
6. History of regular alcohol consumption within 6 months of the study defined as:

   • an average weekly intake of greater than 21 units (14 units for female) or an average daily intake of greater than 3 units (2 units for female). 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
7. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
8. Vulnerable subjects, or subject is mentally or legally incapacitated, or has language barrier precluding adequate understanding of cooperation.
9. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
10. A positive test for HIV antibody.
11. A positive pre-study drug/alcohol screen.
12. Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
13. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
14. Consumption of broccoli, radish sprouts, cauliflower, cabbage, orange juice, apple juice grapefruit juice or grapefruit within 7 days prior to the first dose of study medication until collection of the final pharmacokinetic blood sample.
15. The subject has participated in a clinical trial and has received an investigational product (IP) within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the IP (whichever is longer).
16. Exposure to more than four new chemical entities (i.e., medical drugs being under development) within 12 months prior to the first dosing day.
17. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
18. Unwillingness or inability to follow the procedures outlined in the protocol.
19. The subject is unable or unwilling to abstain from strenuous physical activity in the 48 h before screening and up to the follow up visit.
20. Subject is the investigator or his/her deputies, research assistant, pharmacist, study coordinator, other staff or relative thereof involved in the conduct of the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-01-18 (Actual); Primary Completion 2010-02-26 (Actual); Study Completion 2010-02-26 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability evaluated by adverse event monitoring, ECG, Vital Signs, physical examination, laboratory values and Romberg/heel to toe tests; plasma analysis of Simvastatin and Atorvastatin and active metabolites. | screening period of 28 days followed 17 days clinical duration plus a follow up visit 7-14 days post last dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 109652 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/109652?search=study&search_terms=109652#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 109652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109652 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register